CLINICAL TRIAL: NCT02130986
Title: Procalcitonin Antibiotic Consensus Trial (ProACT)
Acronym: ProACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); BioMérieux (Industry)
Responsible Party: Principal Investigator, David T. Huang, MD, MPH, Associate Professor of Critcal Care and Emergency Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01GM101197 (NIH); 1R01GM101197 (NIH)
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Lower Respiratory Tract Infection (LRTI)
Keywords: procalcitonin (PCT); lower respiratory tract infection (LRTI); antibiotic exposure; antibiotic decision making; community acquired pneumonia (CAP); chronic obstructive pulmonary disease (COPD) exacerbation; acute asthma exacerbation; acute bronchitis; procalcitonin guideline
MeSH Terms: conditions — Community-Acquired Pneumonia; Pulmonary Disease, Chronic Obstructive; Bronchitis | interventions — Procalcitonin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procalcitonin (PCT) group (Experimental): Procalcitonin (PCT) level; Results of procalcitonin level to treating clinician; Provide procalcitonin guideline to treating clinician; Telephone Visit at Day 15 and Day 30
  Interventions: Other: Procalcitonin level; Other: Results of procalcitonin (PCT) level to treating clinician; Other: Provide procalcitonin guideline to treating clinician; Other: Telephone Visit
- Usual Care group (Active Comparator): Telephone Visit at Day 15 and Day 30
  Interventions: Other: Telephone Visit

INTERVENTIONS:
Other: Procalcitonin level — A procalcitonin (PCT) will be drawn level within one hour after randomization in the ED, and if hospitalized, 6-24 hours after the initial ED blood draw, and on Days 3, 5, and 7. Days 3, 5, and 7 blood draws for procalcitonin will only occur in hospitalized patients on antibiotics and/or at the treating physician's discretion.
  Other Names: PCT level
  Arms: Procalcitonin (PCT) group
Other: Results of procalcitonin (PCT) level to treating clinician — In the ED, we will quickly (<1 hour goal) provide clinicians the procalcitonin result.
  Arms: Procalcitonin (PCT) group
Other: Provide procalcitonin guideline to treating clinician — Procalcitonin antibiotic guideline --
  Procalcitonin level (ug/L) -- Bacterial etiology -- Recommendation
  < 0.1 -- Very unlikely -- Antibiotics strongly discouraged(1)
  0.1 - 0.25 -- Unlikely -- Antibiotics discouraged(1)
  > 0.25 - 0.5 -- Likely -- Antibiotics recommended(2)
  > 0.5 -- Very likely -- Antibiotics strongly recommended(2)
  1. Initial antibiotics can be considered for critical illness, Legionella pneumophilia. Procalcitonin should be evaluated in context with all findings and the total clinical status; clinical judgment always necessary.
  2. For outpatients, antibiotic duration based on level (> 0.25-0.5 ug/L:3 days; > 0.5-1.0 ug/L:5 days; >1.0 ug/L:7 days). Physician follow-up is recommended.
  Arms: Procalcitonin (PCT) group
Other: Telephone Visit — We will collect the number of antibiotic days during telephone visits occurring on or around Day 15 and Day 30

SUMMARY:
The ProACT study is a 5 year, multicenter study that will test the effect of implementation of a novel procalcitonin guideline on antibiotic use and adverse outcomes in Emergency Department (ED) patients with Lower Respiratory Tract Infection (LRTI).

DETAILED DESCRIPTION:
There is a need for improved decision-making for antibiotic prescription in acute suspected infection. Infections, particularly in the early stages, can have protean manifestations, often do not manifest with "classic" signs, and clinically overlap with non-infectious conditions. However, the imperative to quickly give antibiotics for bacterial infection has led to antibiotic overuse and resistance.

Strategies that combine novel diagnostics with therapeutics have improved decision-making in oncology, cardiology, and other fields. These strategies aim to identify those patients most likely to be helped or harmed by the therapeutic intervention and allow more individualized care. This approach takes diagnostics to the next level, by demanding a test not only measure well, but also that clinical care be improved by tying the test to a treatment strategy.

Procalcitonin, a novel biomarker of bacterial infection, may help physicians make more appropriate antibiotic decisions. Lower respiratory tract infection (LRTI) is an ideal trial population. LRTI accounts for a large proportion of antibiotic prescription, and exemplifies the imprecise clinical phenotype of infection.However, key questions of generalizability and safety preclude widespread application.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* A primary clinical diagnosis in the ED of acute LRTI (< 28 days duration)
* Clinician willing to consider procalcitonin in antibiotic decision-making

Exclusion Criteria:

* Systemic antibiotics before ED presentation (All prophylactic antibiotic regimens, OR received >1 dose within 72 hours prior to ED presentation)
* Current vasopressor use
* Mechanical ventilation (via endotracheal tube)
* Known severe immunosuppression
* Accompanying non-respiratory infections
* Known lung abscess or empyema
* Chronic dialysis
* Metastatic cancer
* Surgery in the past 7 days (excluding minor surgery such as skin biopsy)
* Incarcerated or homeless
* Enrolled in ProACT in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1664 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Huang, MD MPH, Principal Investigator — University of Pittsburgh
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - University of California at Irvine Medical Center, Orange, California
  - Norwalk Hospital, Norwalk, Connecticut
  - University of Maryland/Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University/Detroit Receiving Hospital, Detroit, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - The Ohio State University, College of Medicine, Columbus, Ohio
  - Penn State Hershey College of Medicine; Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Meisner M. Biomarkers of sepsis: clinically useful? Curr Opin Crit Care. 2005 Oct;11(5):473-80. doi: 10.1097/01.ccx.0000176694.92883.ce. PMID 16175035
- [Background] Schuetz P, Christ-Crain M, Muller B. Procalcitonin and other biomarkers to improve assessment and antibiotic stewardship in infections--hope for hype? Swiss Med Wkly. 2009 Jun 13;139(23-24):318-26. doi: 10.4414/smw.2009.12584. PMID 19529989
- [Background] Muller B, White JC, Nylen ES, Snider RH, Becker KL, Habener JF. Ubiquitous expression of the calcitonin-i gene in multiple tissues in response to sepsis. J Clin Endocrinol Metab. 2001 Jan;86(1):396-404. doi: 10.1210/jcem.86.1.7089. PMID 11232031
- [Background] Nylen E, Muller B, Becker KL, Snider R. The future diagnostic role of procalcitonin levels: the need for improved sensitivity. Clin Infect Dis. 2003 Mar 15;36(6):823-4; author reply 826-7. doi: 10.1086/368088. No abstract available. PMID 12627371
- [Background] Uzzan B, Cohen R, Nicolas P, Cucherat M, Perret GY. Procalcitonin as a diagnostic test for sepsis in critically ill adults and after surgery or trauma: a systematic review and meta-analysis. Crit Care Med. 2006 Jul;34(7):1996-2003. doi: 10.1097/01.CCM.0000226413.54364.36. PMID 16715031
- [Background] Jones AE, Fiechtl JF, Brown MD, Ballew JJ, Kline JA. Procalcitonin test in the diagnosis of bacteremia: a meta-analysis. Ann Emerg Med. 2007 Jul;50(1):34-41. doi: 10.1016/j.annemergmed.2006.10.020. Epub 2006 Dec 11. PMID 17161501
- [Background] Simon L, Gauvin F, Amre DK, Saint-Louis P, Lacroix J. Serum procalcitonin and C-reactive protein levels as markers of bacterial infection: a systematic review and meta-analysis. Clin Infect Dis. 2004 Jul 15;39(2):206-17. doi: 10.1086/421997. Epub 2004 Jul 2. PMID 15307030
- [Background] Stolz D, Christ-Crain M, Gencay MM, Bingisser R, Huber PR, Muller B, Tamm M. Diagnostic value of signs, symptoms and laboratory values in lower respiratory tract infection. Swiss Med Wkly. 2006 Jul 8;136(27-28):434-40. doi: 10.4414/smw.2006.11271. PMID 16862463
- [Background] Hirakata Y, Yanagihara K, Kurihara S, Izumikawa K, Seki M, Miyazaki Y, Kohno S. Comparison of usefulness of plasma procalcitonin and C-reactive protein measurements for estimation of severity in adults with community-acquired pneumonia. Diagn Microbiol Infect Dis. 2008 Jun;61(2):170-4. doi: 10.1016/j.diagmicrobio.2008.01.014. Epub 2008 Mar 7. PMID 18329217
- [Background] Prieto B, Llorente E, Gonzalez-Pinto I, Alvarez FV. Plasma procalcitonin measured by time-resolved amplified cryptate emission (TRACE) in liver transplant patients. A prognosis marker of early infectious and non-infectious postoperative complications. Clin Chem Lab Med. 2008;46(5):660-6. doi: 10.1515/cclm.2008.123. PMID 18839468
- [Background] Prat C, Sancho JM, Dominguez J, Xicoy B, Gimenez M, Ferra C, Blanco S, Lacoma A, Ribera JM, Ausina V. Evaluation of procalcitonin, neopterin, C-reactive protein, IL-6 and IL-8 as a diagnostic marker of infection in patients with febrile neutropenia. Leuk Lymphoma. 2008 Sep;49(9):1752-61. doi: 10.1080/10428190802258956. PMID 18661397
- [Background] Charles PE, Kus E, Aho S, Prin S, Doise JM, Olsson NO, Blettery B, Quenot JP. Serum procalcitonin for the early recognition of nosocomial infection in the critically ill patients: a preliminary report. BMC Infect Dis. 2009 Apr 22;9:49. doi: 10.1186/1471-2334-9-49. PMID 19386110
- [Background] Huang DT, Weissfeld LA, Kellum JA, Yealy DM, Kong L, Martino M, Angus DC; GenIMS Investigators. Risk prediction with procalcitonin and clinical rules in community-acquired pneumonia. Ann Emerg Med. 2008 Jul;52(1):48-58.e2. doi: 10.1016/j.annemergmed.2008.01.003. Epub 2008 Mar 17. PMID 18342993
- [Background] Muller B, Harbarth S, Stolz D, Bingisser R, Mueller C, Leuppi J, Nusbaumer C, Tamm M, Christ-Crain M. Diagnostic and prognostic accuracy of clinical and laboratory parameters in community-acquired pneumonia. BMC Infect Dis. 2007 Mar 2;7:10. doi: 10.1186/1471-2334-7-10. PMID 17335562
- [Background] Cuquemelle E, Soulis F, Villers D, Roche-Campo F, Ara Somohano C, Fartoukh M, Kouatchet A, Mourvillier B, Dellamonica J, Picard W, Schmidt M, Boulain T, Brun-Buisson C; A/H1N1 REVA-SRLF Study Group. Can procalcitonin help identify associated bacterial infection in patients with severe influenza pneumonia? A multicentre study. Intensive Care Med. 2011 May;37(5):796-800. doi: 10.1007/s00134-011-2189-1. Epub 2011 Mar 3. PMID 21369807
- [Background] Schappert SM, Rechtsteiner EA. Ambulatory medical care utilization estimates for 2007. Vital Health Stat 13. 2011 Apr;(169):1-38. PMID 21614897
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Stolz D, Christ-Crain M, Bingisser R, Leuppi J, Miedinger D, Muller C, Huber P, Muller B, Tamm M. Antibiotic treatment of exacerbations of COPD: a randomized, controlled trial comparing procalcitonin-guidance with standard therapy. Chest. 2007 Jan;131(1):9-19. doi: 10.1378/chest.06-1500. PMID 17218551
- [Background] Schuetz P, Christ-Crain M, Thomann R, Falconnier C, Wolbers M, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Regez K, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Effect of procalcitonin-based guidelines vs standard guidelines on antibiotic use in lower respiratory tract infections: the ProHOSP randomized controlled trial. JAMA. 2009 Sep 9;302(10):1059-66. doi: 10.1001/jama.2009.1297. PMID 19738090
- [Background] Long W, Deng X, Zhang Y, Lu G, Xie J, Tang J. Procalcitonin guidance for reduction of antibiotic use in low-risk outpatients with community-acquired pneumonia. Respirology. 2011 Jul;16(5):819-24. doi: 10.1111/j.1440-1843.2011.01978.x. PMID 21507143
- [Derived] Malley BE, Yabes JG, Gimbel E, Chang CH, Yealy DM, Fine MJ, Angus DC, Huang DT; ProACT Investigators. Impact of adherence to procalcitonin antibiotic prescribing guideline recommendations for low procalcitonin levels on antibiotic use. BMC Infect Dis. 2023 Jan 19;23(1):30. doi: 10.1186/s12879-022-07923-0. PMID 36658543
- [Derived] Huang DT, Yealy DM, Filbin MR, Brown AM, Chang CH, Doi Y, Donnino MW, Fine J, Fine MJ, Fischer MA, Holst JM, Hou PC, Kellum JA, Khan F, Kurz MC, Lotfipour S, LoVecchio F, Peck-Palmer OM, Pike F, Prunty H, Sherwin RL, Southerland L, Terndrup T, Weissfeld LA, Yabes J, Angus DC; ProACT Investigators. Procalcitonin-Guided Use of Antibiotics for Lower Respiratory Tract Infection. N Engl J Med. 2018 Jul 19;379(3):236-249. doi: 10.1056/NEJMoa1802670. Epub 2018 May 20. PMID 29781385
- [Derived] Huang DT, Angus DC, Chang CH, Doi Y, Fine MJ, Kellum JA, Peck-Palmer OM, Pike F, Weissfeld LA, Yabes J, Yealy DM; ProACT Investigators. Design and rationale of the Procalcitonin Antibiotic Consensus Trial (ProACT), a multicenter randomized trial of procalcitonin antibiotic guidance in lower respiratory tract infection. BMC Emerg Med. 2017 Aug 29;17(1):25. doi: 10.1186/s12873-017-0138-1. PMID 28851296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the Emergency Department (ED) if they had a primary clinical diagnosis of acute Lower Respiratory Tract Infection [LRTI] (< 28 days duration) and their key clinician was willing to consider Procalcitonin (PCT) result in Antibiotic (ABX) decision making.
Pre-assignment Details: Only 8 patients (4 in each arm) were entirely excluded because they withdrew all consent to participate.
Groups:
- Procalcitonin (PCT) Group: Procalcitonin (PCT)
  Results of procalcitonin level provided to treating clinician (initial in the ED, 6-24 hrs after initial. and Day 3, 5, 7 if in hospital AND on abx or at the treating clinician's discretion)
  Telephone Visit at Day 15 and Day 30 to collect ABX days, post-d/c resource use and AQ-20 questionnaire
  Bio-bank samples collected in ED for storage at Coordinating Center
- Usual Care (UC) Group: Usual Care
  Telephone Visit at Day 15 and Day 30 to collect ABX days, post-d/c resource use and AQ-20 questionnaire
  Bio-bank samples collected in ED for storage at Coordinating Center
Period: Overall Study
Arm/Group | Procalcitonin (PCT) Group | Usual Care (UC) Group
Started | 830 | 834
Completed | 675 | 670
Not Completed | 155 | 164
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 151 | 160

BASELINE CHARACTERISTICS:
Population: Only excluded 4 patients in each group for a total of 8 subjects. These 8 subjects withdrew all consent for participation.
Groups:
- Procalcitonin (PCT) Group: Procalcitonin level: A procalcitonin (PCT) will be drawn level within one hour after randomization in the ED, and if hospitalized, 6-24 hours after the initial ED blood draw, and on Days 3, 5, and 7. Days 3, 5, and 7 blood draws for procalcitonin will only occur in hospitalized patients on antibiotics and/or at the treating physician's discretion.
  Results of procalcitonin (PCT) level to treating clinician: In the ED, we will quickly (<1 hour goal) provide clinicians the procalcitonin result.
  Provide PCT guideline to treating clinician: Procalcitonin antibiotic guideline --
  PCT level (ug/L)-- Bacterial etiology -- Recommendation < 0.1-- Very unlikely -- Antibiotics strongly discouraged 0.1 - 0.25 -- Unlikely--Antibiotics discouraged > 0.25 - 0.5--Likely -- Antibiotics recommended > 0.5-- Very likely -- Antibiotics strongly recommended
  Telephone Visit: We will collect the number of antibiotic days during telephone visits occurring on or around Day 15 and Day 30
- Usual Care (UC) Group: Telephone Visit at Day 15 and Day 30
  Telephone Visit: We will collect the number of antibiotic days during telephone visits occurring on or around Day 15 and Day 30
- Total: Total of all reporting groups
Arm/Group | Procalcitonin (PCT) Group | Usual Care (UC) Group | Total
Number analyzed (Participants) | 826 | 830 | 1656
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 7 | 12
  Between 18 and 65 years | 603 | 596 | 1199
  >=65 years | 218 | 227 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (18.4) | 53.2 (18.7) | 53.1 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 469 | 476 | 945
  Male | 357 | 354 | 711
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 455 | 470 | 925
  Black | 296 | 297 | 593
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was self-reported and information was requested prior to race description Population: Race and ethnic group were reported by the patients.
  Participants
    Hispanic: number analyzed (Participants) | 815 | 812 | 1627
    Hispanic | 108 | 104 | 212
Region of Enrollment [Number; unit: participants]
  United States | 826 | 830 | 1656

OUTCOME MEASURES:

1. Primary Outcome: Total Antibiotic Exposure Days
Description: Total antibiotic exposure, defined as the total number of antibiotic-days by Day 30.
Time Frame: 30 days
Population: Mixed modeling was used to impute missing data for the intention-to-treat analysis for the primary outcome since not all patients could be reached for the 30 day interview (which collected 30 day antibiotic use).
Measure: Mean (Standard Deviation); unit: days
Groups:
- Procalcitonin (PCT) Group: Procalcitonin (PCT) level; Results of procalcitonin level to treating clinician; Provide procalcitonin guideline to treating clinician; Telephone Visit at Day 15 and Day 30
  Procalcitonin level: A procalcitonin (PCT) will be drawn level within one hour after randomization in the ED, and if hospitalized, 6-24 hours after the initial ED blood draw, and on Days 3, 5, and 7. Days 3, 5, and 7 blood draws for procalcitonin will only occur in hospitalized patients on antibiotics and/or at the treating physician's discretion.
  Results of procalcitonin (PCT) level to treating clinician: In the ED, we will quickly (<1 hour goal) provide clinicians the procalcitonin result.
  Provide procalcitonin guideline to treating clinician.
Arm/Group | Procalcitonin (PCT) Group | Usual Care Group
Number analyzed (Participants) | 826 | 830
days | 4.2 (5.8) | 4.3 (5.6)
Statistical Analysis 1: Comparison: Procalcitonin (PCT) Group vs Usual Care Group; Test type: Superiority; p = 0.87, t-test, 2 sided; Mean Difference (Net) = -0.05

2. Primary Outcome: Number of Participants With Any Adverse Outcome
Description: Primary Safety Outcome - Combined endpoint of adverse outcomes (death, endotracheal intubation, vasopressors, renal failure, lung abscess/empyema, pneumonia in non-CAP patient, and hospital readmissions) that could be attributable to withholding antibiotics in lower respiratory tract infection (LRTI).
  Number is based on the number of participants that experienced any adverse outcome.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Procalcitonin (PCT) Group: Provide PCT results and procalcitonin guideline to treating clinician; Telephone Visit at Day 15 and Day 30 for # of ABX days
  A procalcitonin (PCT) will be drawn within one hour after randomization in the ED, and if hospitalized, 6-24 hours after the initial ED blood draw, and on Days 3, 5, and 7. Days 3, 5, and 7 blood draws for procalcitonin will only occur in hospitalized patients on antibiotics and/or at the treating physician's discretion. Results & guideline provided to the treating clinician.
  PCT guideline to treating clinician:
  Procalcitonin level (ug/L) -- Bacterial etiology -- Recommendation
  < 0.1 --Very unlikely -- Antibiotics strongly discouraged
  0.1 - 0.25 -- Unlikely --Antibiotics discouraged
  > 0.25 -- 0.5--Likely--Antibiotics recommended
  > 0.5 --Very likely -- Antibiotics strongly recommended
Arm/Group | Procalcitonin (PCT) Group | Usual Care Group
Number analyzed (Participants) | 826 | 830
Participants | 96 | 109
Statistical Analysis 1: Comparison: Procalcitonin (PCT) Group vs Usual Care Group; Test type: Non-Inferiority — Procalcitonin algorithm implementation increases or does not change the proportion of subjects who experience a composite endpoint of adverse outcomes by Day 30. The prespecified noninferiority margin is 4.5 percentage; p < 0.001, Chi-squared; Risk Difference (RD) = -0.015

3. Secondary Outcome: Antibiotic Prescription in Emergency Department(ED)
Description: Antibiotic prescription in the ED includes post-randomization receipt of antibiotics in ED and provision of an antibiotic prescription for patients at the time of discharge from the ED.
Time Frame: While in the ED or before ED discharge (majority patients < 1 day)
Measure: Count of Participants; unit: Participants
Groups:
- Procalcitonin (PCT) Group: Procalcitonin (PCT) level; Results of procalcitonin level to treating clinician; Provide procalcitonin guideline to treating clinician; Telephone Visit at Day 15 and Day 30
  Procalcitonin level: A procalcitonin (PCT) will be drawn level within one hour after randomization in the ED, and if hospitalized, 6-24 hours after the initial ED blood draw, and on Days 3, 5, and 7. Days 3, 5, and 7 blood draws for procalcitonin will only occur in hospitalized patients on antibiotics and/or at the treating physician's discretion.
  Results of procalcitonin (PCT) level to treating clinician: In the ED, we will quickly (<1 hour goal) provide clinicians the procalcitonin result.
  Provide procalcitonin guideline to treating clinician: Procalcitonin antibiotic guideline --
  Procalcitonin level (ug/L) -- Bacterial etiology -- Recommendation < 0.1 -- Very unlikely -- Antibiotics strongly discouraged(1) 0.1 - 0.25 -- Unlikely -- Antibiotics discouraged(1
Arm/Group | Procalcitonin (PCT) Group | Usual Care Group
Number analyzed (Participants) | 826 | 830
Participants | 282 | 321
Statistical Analysis 1: Comparison: Procalcitonin (PCT) Group vs Usual Care Group; Test type: Superiority; Risk Difference (RD) = -4.6, 95% CI 2-sided [-12.2 to 30]

ADVERSE EVENTS:
Time Frame: By day 30.
Description: All events were reviewed and assessed by the Principal Investigator at the participating site.
  8 patients (4 in each arm) were entirely excluded because they withdrew all consent to participate.
  Most specific terms are reported in the Adverse Event Section.
Groups:
- Usual Care Group: Usual Care
  Telephone Visit at Day 15 and Day 30 to collect ABX days, post-d/c resource use and AQ-20 questionnaire
  Bio-bank samples collected in ED for storage at Coordinating Center
Arm/Group | Procalcitonin (PCT) Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 16/826 | 10/830
Serious Adverse Events (participants affected / at risk) | 14/826 | 9/830
Other Adverse Events (participants affected / at risk) | 20/826 | 14/830
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procalcitonin (PCT) Group (N=826) | Usual Care Group (N=830)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Death NOS (General disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient developed pseudomonas PNA while in hospital
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procalcitonin (PCT) Group (N=826) | Usual Care Group (N=830)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — No descriptions
Death NOS (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT02130986/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02130986/SAP_001.pdf